CLINICAL TRIAL: NCT02729116
Title: Sitafloxacin and Ertapenem Treatment for Acute Urinary Tract Infection Caused by E. Coli or K. Pneumoniae in Post-kidney Transplantation Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Atibordee Meesing, MD, Principal Investigator, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HE581520
Record Dates: First submitted 2016-03-24; First posted 2016-04-06 (Estimated); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Anti-Infective Agents, Urinary; Escherichia Coli Infections; Klebsiella Infections; Kidney Transplantation; Urinary Tract Infections
Keywords: Extended-Spectrum ß-lactamase-producing Escherichia coli; Extended-Spectrum ß-lactamase-producing Klebsiella pneumoniae; Kidney Transplantation; Urinary Tract Infections
MeSH Terms: conditions — Escherichia coli Infections; Klebsiella Infections; Urinary Tract Infections | interventions — sitafloxacin; Ertapenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sitafloxacin group (Experimental): Sitafloxacin 100 mg oral twice daily
  Interventions: Drug: Sitafloxacin
- Ertapenem group (Active Comparator): Ertapenem 1 gm IV every 24 h
  Interventions: Drug: Ertapenem

INTERVENTIONS:
Drug: Sitafloxacin — Patients are given intravenous empirical antibiotics for 3 days. The patients are allocated to the sitafloxacin group or ertapenem group using of a computer-generated random number allocation schedule and block size of four.
  Arms: Sitafloxacin group
Drug: Ertapenem — Patients are given IV ertapenem for 14 days
  Arms: Ertapenem group

SUMMARY:
This study evaluates oral antimicrobial agents for the treatment of non-bacteremic acute urinary tract infection caused by Extended Spectrum Beta Lactamase producing Escherichia coli or Klebsiella pneumoniae in Post-kidney transplantation. Patients are treated with intravenous (IV) antibiotics follow by oral sitafloxacin or IV ertapenem.

DETAILED DESCRIPTION:
A prospective randomized controlled trial of patients with a presumptive diagnosis of acute urinary tract infection caused by Extended Spectrum Beta Lactamase-producing Escherichia coli or Klebsiella pneumoniae in Post-kidney transplantation. Intravenous (IV) antibiotic is initially given to all patients. After day 3, patients were randomized to receive either oral sitafloxacin (100 mg twice daily) or intravenous ertapenem. The course of treatment will complete within 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Acute urinary infection by definitions
* Positive urine culture for Extended Spectrum Beta Lactamase E. coli or K. pneumoniae ≥105 colony forming unit/mL
* Post-kidney transplantation
* Voluntarily consented to be enrolled in the study

Exclusion Criteria:

* Sepsis
* Positive blood culture
* Mixed organism of urine culture
* Immunocompromised conditions other than post-kidney transplantation
* Pregnancy or lactation
* Previous urinary tract infections within 4 weeks
* Contraindicated for fluoroquinolones and carbapenems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with clinical cure of acute urinary tract infection | 14 days
  No symptoms of acute urinary tract infection

SECONDARY OUTCOMES:
Number of patients with micrological cure of acute urinary tract infection | 14 days
  No evidence of Extended Spectrum Beta Lactamase Escherichia coli or Klebsiella pneumoniae in urine culture

CONTACTS AND LOCATIONS:
Locations (1):
- Khon Kaen University, Ban Khanaen, Khonkaen, Thailand

REFERENCES:
- [Background] Thamlikitkul V, Tiengrim S. In vitro susceptibility test of sitafloxacin against resistant gram-negative bacilli isolated from Thai patients by disk diffusion method. J Med Assoc Thai. 2014 Mar;97 Suppl 3:S7-12. PMID 24772575
- [Background] Nakamura T, Komatsu M, Yamasaki K, Fukuda S, Higuchi T, Ono T, Nishio H, Sueyoshi N, Kida K, Satoh K, Toda H, Toyokawa M, Nishi I, Sakamoto M, Akagi M, Mizutani T, Nakai I, Kofuku T, Orita T, Zikimoto T, Natsume S, Wada Y. Susceptibility of various oral antibacterial agents against extended spectrum beta-lactamase producing Escherichia coli and Klebsiella pneumoniae. J Infect Chemother. 2014 Jan;20(1):48-51. doi: 10.1016/j.jiac.2013.08.004. Epub 2013 Dec 11. PMID 24462425
- [Background] Tiengrim S, Phiboonbanakit D, Thunyaharn S, Tantisiriwat W, Santiwatanakul S, Susaengrat W, Srisurat N, Malithong A, Srisangchan P, Thamlikitkul V. Comparative in vitro activity of sitafloxacin against bacteria isolated from Thai patients with urinary tract infections and lower respiratory tract infections. J Med Assoc Thai. 2012 Feb;95 Suppl 2:S6-17. PMID 22574524